CLINICAL TRIAL: NCT00832416
Title: A Four-Arm Study Comparing the Analgesic Efficacy and Safety of Tramadol Once a Day 100, 200 and 300 mg Versus Placebo for the Treatment of Pain Due to Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDT3-002; NCT00832416 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Pain; Osteoarthritis, Knee
MeSH Terms: conditions — Pain; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 Tramadol Once A Day 100mg (Experimental)
  Interventions: Drug: Tramadol Once A Day
- 2: Tramadol Once A Day 200mg (Experimental)
  Interventions: Drug: Tramadol Once A Day
- 3: Tramadol Once A Day 300mg (Experimental)
  Interventions: Drug: Tramadol Once A Day
- 4: Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol Once A Day — One Tramadol Once A Day tablet at randomized dose daily.
  Arms: 1 Tramadol Once A Day 100mg; 2: Tramadol Once A Day 200mg; 3: Tramadol Once A Day 300mg
Drug: Placebo — One Placebo tablet daily.
  Arms: 4: Placebo

SUMMARY:
The purpose of this study is to compare the analgesic efficacy and safety of Tramadol Once a Day 100, 200, 300 mg and Placebo

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females between the ages of 40-75 with a diagnosis of moderate to severe osteoarthritis of the knee, consistent with the American College of Rheumatology (ACR) Clinical Classification Criteria for Arthritis of the Knee:

   * Current knee pain
   * Less than 30 minutes of morning stiffness with or without crepitus on active motion.
   * Confirmation either by arthroscopy or radiologist's report (X-rays showing osteophytes, joint space narrowing or subchondral bone sclerosis {eburnation}) within five years prior to entry into the study.
2. C-reactive protein (CRP) < 8 ug/ml (if available at local lab) or erythrocyte sedimentation rate (ESR) < 40 mm/hr
3. Total WOMAC (Western Ontario and McMaster University Osteoarthritis Index) Pain Subscale Score of > 150 mm at Baseline corresponding with moderate to severe Osteoarthritis.
4. Oral and written language comprehension at a level sufficient to comply with the protocol and complete study-related materials.
5. Research Ethics Board (REB) approval of the written Informed Consent Form in Spanish or English which was signed and dated by the patient and Investigator, prior to study participation.

Exclusion Criteria:

1. Known rheumatoid arthritis or any other rheumatoid disease.
2. Secondary arthritis i.e. any of the following: septic arthritis; inflammatory joint disease; gout; pseudogout; Paget's disease; joint fracture; acromegaly; fibromyalgia; Wilson's disease; ochronosis; haemochromatosis; osteochondromatosis; or collagen gene mutations.
3. Evidence of effusion greater than 15 cubic centimetre (cc) upon physical examination of the joint at Baseline (Visit 1).
4. Body Mass Index (BMI) ≥ 38.
5. Major illness, requiring hospitalization during the 3 months before commencement of the screening period.
6. The patient was unwilling to stop taking pain medication (for arthritis or other types of pain) or was unwilling to stop taking other medications for the treatment of osteoarthritis (OA).
7. Previous failure or discontinuation (due to adverse events) of tramadol hydrochloride (HCl) therapy.
8. Treatment within the last 3 weeks with any of the following medications: monoamine oxidase inhibitors; tricyclic antidepressants and other tricyclic compounds (e.g. cyclobenzaprine, promethazine); neuroleptics; selective serotonin reuptake inhibitors; or any other drug that reduces seizure threshold.
9. Treatment with another investigational agent within the last 30 days.
10. A history of seizure disorder other than Infantile Febrile Seizures.
11. Previous or current opioid dependency.
12. Bowel disease causing malabsorption.
13. Pregnancy or lactating or childbearing potential and unwilling to utilize a medically approved method of contraception during participation in this clinical trial.
14. Significant liver disease, defined as active hepatitis or elevated liver enzymes >3 times the upper boundary of the normal range.
15. Significant renal disease, defined as creatinine clearance <30 mL/min as estimated by the method of Levey et al., 1999.
16. Current substance abuse or dependence, other than nicotine.
17. Allergy or adverse reaction to tramadol or any structurally similar drugs e.g. opiates.
18. Any other condition, that, in the opinion of the Investigators, would have adversely affected the patient's ability to complete the study or its measures.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2003-01; Primary Completion 2003-08 (Actual)

REFERENCES:
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=9048

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Started | 110 | 113 | 115 | 227
Completed | 64 | 60 | 54 | 144
Not Completed | 46 | 53 | 61 | 83
Not completed — Lack of Efficacy | 17 | 15 | 13 | 52
Not completed — Withdrawal by Subject | 5 | 7 | 2 | 10
Not completed — Physician Decision | 2 | 12 | 5 | 10
Not completed — Administrative | 0 | 0 | 0 | 1
Not completed — Adverse Event | 21 | 19 | 41 | 10
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo | Total
Number analyzed (Participants) | 110 | 113 | 115 | 227 | 565
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 69 | 77 | 66 | 139 | 351.0
  >=65 years | 41 | 36 | 49 | 88 | 214.0
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.0) | 59.8 (8.4) | 61.0 (9.6) | 60.6 (9.6) | 60.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 72 | 140 | 341.0
  Male | 45 | 49 | 43 | 87 | 224.0

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Rating of Pain for the Study Period (12 Weeks)
Description: 3-item Likert-scale: "How do you rate overall pain relief with the drug?" with 3 possible answers: "very effective", "effective", or "ineffective". The average of ratings at visits 2-5 was calculated as median, rounded up to the closest integer.
Time Frame: 12 weeks
Population: The analysis was performed using the full analysis population (All randomized patients who received at least one dose of the assigned study medication and had at least one post Baseline assessment of any functional scale). Last Individual value.
Measure: Number; unit: participants
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 108 | 109 | 113 | 223
participants
  Very effective | 19 | 16 | 26 | 29
  Effective | 50 | 56 | 56 | 94
  Ineffective | 39 | 37 | 31 | 100

2. Primary Outcome: Percentage Difference Between WOMAC Pain Subscale Score From Baseline to the End of the Study (Week 12)
Description: Percentage of difference in WOMAC Pain Subscale score between baseline and week 12. The WOMAC scale is a 24-item questionnaire divided in 3 subscales, using a 100mm visual analog scale ranging from no pain (0mm) to extreme pain (100mm). The WOMAC Pain Subscale results from the sum of 5 questions.
Time Frame: Baseline to week 12
Population: The analysis was performed using the full analysis population (All randomized patients who received at least one dose of the assigned study medication and had at least one post Baseline assessment of any functional scale). Missing Values at Last Visit Imputed by Individual Last Post Baseline Value.
Measure: Mean (Standard Deviation); unit: Percentage difference
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 109 | 110 | 113 | 226
Percentage difference | 36.3 (45.3) | 36.6 (40.9) | 41.0 (44.5) | 38.0 (41.7)

3. Secondary Outcome: Percentage Difference in WOMAC Pain Subscale Score From Baseline to Intervening Visits (Visits 2-4)
Description: Percentage of difference in WOMAC Pain Subscale score between baseline and intervening visits 2-4. The WOMAC scale is a 24-item questionnaire divided in 3 subscales, using a 100mm visual analog scale ranging from no pain (0mm) to extreme pain (100mm). The WOMAC Pain Subscale results from the sum of 5 questions.
Time Frame: Week 0, week 3, week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage difference
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 109 | 110 | 113 | 226
Percentage difference
  Week 0 (Visit 2) | 26.7 (36.9) | 29.0 (33.4) | 33.1 (41.4) | 20.4 (35.8)
  Week 3 (Visit 3) | 35.2 (40.9) | 36.0 (40.3) | 42.3 (40.6) | 35.1 (39.4)
  Week 6 (Visit 4) | 36.3 (40.9) | 36.4 (39.5) | 47.7 (42.2) | 41.3 (39.9)

4. Secondary Outcome: Percentage Difference in WOMAC Physical Function Subscale Score From Baseline to Intervening Visits (Visits 2-4)
Description: Percentage of difference in WOMAC Physical Function Subscale score between baseline and intervening visits 2-4. The WOMAC scale is a 24-item questionnaire divided in 3 subscales. The WOMAC Physical Function Subscale comprises 17 questions each rated on a 100mm visual analog scale (VAS) ranging from no pain (0mm) to extreme pain (100mm).
Time Frame: Week 0, week 3, week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage difference
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 109 | 110 | 113 | 226
Percentage difference
  Week 0 (Visit 2) | 23.4 (37.1) | 26.4 (30.9) | 29.3 (37.9) | 18.5 (37.7)
  Week 3 (Visit 3) | 33.3 (40.7) | 36.5 (34.4) | 41.0 (39.7) | 33.7 (38.2)
  Week 6 (Visit 4) | 33.5 (39.8) | 37.0 (36.8) | 47.7 (43.8) | 38.3 (37.8)

5. Secondary Outcome: Multiple Dose Effect Using 24-hour VAS Pain Questionnaire
Description: Patients rated their knee pain by marking a 100mm Visual Analogue Scale, ranging from no pain (0mm) to extreme pain (100mm).
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 109 | 110 | 113 | 226
mm
  Pain at lunchtime (last individual visit) | 40.5 (29.9) | 38.2 (29.6) | 36.6 (29.4) | 38.5 (29.5)
  Pain at bed time (last individual visit) | 41.2 (30.7) | 41.1 (29.9) | 37.3 (30.2) | 39.7 (29.4)
  Pain Before next morning dose (last individ visit) | 41.1 (30.1) | 42.0 (29.5) | 35.5 (29.3) | 38.5 (29.8)

6. Secondary Outcome: Investigator Global Rating of Pain Relief
Description: The Investigator Global Rating of Pain is a 3-item Likert-scale to answer the following question: "How do you rate this patient's overall pain relief with the drug?" with 3 possible answers: "very effective", "effective", or "ineffective".
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 108 | 109 | 111 | 223
participants
  Very effective | 20 | 14 | 22 | 29
  Effective | 49 | 58 | 57 | 98
  Ineffective | 39 | 37 | 32 | 96

7. Primary Outcome: Percentage Difference Between WOMAC Physical Function Subscale Score From Baseline to the End of the Study (Week 12)
Description: Percentage of difference in WOMAC Physical Function Subscale score between baseline and week 12. The WOMAC scale is a 24-item questionnaire divided in 3 subscales, using a 100mm visual analog scale ranging from no pain (0mm) to extreme pain (100mm). The WOMAC Physical Function subscale results from the sum of 17 questions.
Time Frame: Baseline to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage difference
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 109 | 110 | 113 | 226
Percentage difference | 31.9 (46.0) | 37.0 (39.3) | 37.3 (41.7) | 33.7 (44.3)

8. Secondary Outcome: Percentage of Participants Who Dropped Out From Trial by Dropout Reason
Description: Reasons for withdrawal from the trial were collected and the percentage of participants who dropped out from trial were calculated by dropout reason
Time Frame: 12 weeks
Population: Safety population: all randomized patients who received at least one dose of the assigned study medication.
Measure: Number; unit: percentage of participants
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Number analyzed (Participants) | 110 | 113 | 115 | 227
percentage of participants
  Lack of efficacy | 15.5 | 13.3 | 11.3 | 22.9
  Patient request | 4.5 | 6.2 | 1.7 | 4.4
  Investigator initiated discontinuation | 1.8 | 10.6 | 4.3 | 4.4
  Administrative | 0 | 0 | 0 | 0.4
  Adverse event | 19.1 | 16.8 | 35.7 | 4.4
  Death | 0.9 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 1: Tramadol Once A Day 100mg | 2: Tramadol Once A Day 200mg | 3: Tramadol Once A Day 300mg | 4: Placebo
Serious Adverse Events (participants affected / at risk) | 2/110 | 1/113 | 4/115 | 3/227
Other Adverse Events (participants affected / at risk) | 31/110 | 49/113 | 57/115 | 38/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Tramadol Once A Day 100mg (N=110) | 2: Tramadol Once A Day 200mg (N=113) | 3: Tramadol Once A Day 300mg (N=115) | 4: Placebo (N=227)
Bipolar disorder NEC (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep venous thrombosis NOS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer invasive NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis aggravated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecal impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis NOS limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Tramadol Once A Day 100mg (N=110) | 2: Tramadol Once A Day 200mg (N=113) | 3: Tramadol Once A Day 300mg (N=115) | 4: Placebo (N=227)
Constipation (Gastrointestinal disorders) | 10 (10) | 17 (20) | 18 (20) | 15 (17)
Dizziness (Nervous system disorders) | 7 (7) | 20 (20) | 25 (33) | 5 (6)
Nausea (Nervous system disorders) | 17 (18) | 25 (29) | 32 (39) | 14 (14)
Vomiting (Gastrointestinal disorders) | 4 (4) | 8 (9) | 14 (18) | 2 (2)
Headache (Nervous system disorders) | 7 (8) | 6 (12) | 10 (12) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting results communications, the investigator shall allow Labopharm at least 30 days to review the proposed communication. If the proposed publication/disclosure risks Labopharm's ability to patent any invention related to the study, the publication or disclosure will be modified or delayed to allow Labopharm to seek patent protection. This statement does not give Labopharm any editorial rights other than to restrict the disclosure of Labopharm's confidential information.